CLINICAL TRIAL: NCT02309541
Title: Evaluation of a New Feedback Canceller Algorithm for Patient With Moderate to Severe Hearing Loss Implanted With a Fully Implantable Carina™ Medical Device
Brief Title: Evaluation of New Feedback Canceller for Carina™ Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CFRA-A01/CEL5584
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Hearing Loss
Keywords: middle ear implant; feedback manager; Sound quality
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Firmware N (Experimental): New feedback canceller algorithm
  Interventions: Device: feedback canceller algorithm (Firmware)
- Firmware R (Active Comparator): Current feedback canceller algorithm (reference)
  Interventions: Device: feedback canceller algorithm (Firmware)

INTERVENTIONS:
Device: feedback canceller algorithm (Firmware) — The study consists of two phases. Phase 1: optimization of parameters of new feedback canceller algorithm. Phase 2: comparison of new and reference feedback canceller algorithms.

SUMMARY:
The purpose of this study is to evaluate audio quality benefit for the patient implanted with a Cochlear or Otologics Carina implant with the new firmware (feedback canceller algorithm) whatever the patient environment is and to evaluate the functional gain and speech understanding benefit for the patient upon the firmware used (new and reference firmware). The new firmware aims to adapt automatically for feedback cancellation without prior calibration.

ELIGIBILITY:
Inclusion Criteria:

* successfully implanted with a commercial available CE-labelled implant device, resulting in measurable open set speech understanding
* native speaker in the language used to assess their clinical performance, i.e. French

Exclusion Criteria:

* unwillingness or inability to comply with all of the investigational requirements
* additional handicaps that would prevent or restrict participation in the audiological evaluations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Sound quality benefit assessed via subjective patient evaluation with Abbreviated Profile of Hearing Aid Benefit questionnaire | 1 month
Sound quality benefit assessed via subjective patient evaluation with Abbreviated Profile of Hearing Aid Benefit questionnaire | 2 months
Sound quality benefit assessed via subjective patient evaluation with Abbreviated Profile of Hearing Aid Benefit questionnaire | 3 months
Sound quality benefit assessed via subjective patient evaluation with Abbreviated Profile of Hearing Aid Benefit questionnaire | 4 months

SECONDARY OUTCOMES:
Improvement in speech understanding assessed via speech audiometry in noise | 1 month
Improvement in speech understanding assessed via speech audiometry in noise | 2 months
Improvement in speech understanding assessed via speech audiometry in noise | 3 months
Improvement in speech understanding assessed via speech audiometry in noise | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Tringali, Prof, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hôpital Nord, Marseille, Bouches-du-Rhône
  - Hôpital Edouard Herriot, Lyon, Rhône
  - CHU Lyon Sud, Pierre-Bénite, Rhône